CLINICAL TRIAL: NCT01335529
Title: Pilot Study to Assess the Efficacy and Safety of Boceprevir, in Combination With Peg-Interferon Alfa and Ribavirin, in Patients With HCV/HIV Co-infection Who Have Failed to a Previous Therapy With Peg-Interferon/Ribavirin
Brief Title: Boceprevir in HIV-HCV Coinfected Patients Who Have Failed to a Previous Therapy With Peg-Interferon/Ribavirin
Acronym: BocepreVIH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Rennes University Hospital (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS HC27 BOCEPREVIH
Record Dates: First submitted 2011-03-25; First posted 2011-04-14 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: HCV Coinfection; HIV-1 Infection
Keywords: HCV infection; HIV-1 infection
MeSH Terms: conditions — Hepatitis C | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; Ribavirin; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Boceprevir, PegIFN alfa 2b, Ribavirin (Experimental): Standard Treatment :
  * Peg-Interferon (PegIFN) alfa 2b by subcutaneous injection 1,5 µg/kg/week
  * Ribavirin capsules 200mg: dosage delivered in weight categories (< 65 kg: 800 mg ; 65-80 kg: 1000 mg; 81-105 kg: 1200mg; > 105 kg: 1400mg)
  Three-drug-regimen:
  * Peg-Interferon alfa 2b by subcutaneous injection 1,5 µg/kg/week
  * Ribavirin capsules 200mg: dosage delivered in weight categories like in standard treatment
  * Boceprevir tablets 200mg: 800 mg 3 times a day (2400 mg/j) with food
  Interventions: Drug: Boceprevir, Peg-interferon alfa 2b and Ribavirin

INTERVENTIONS:
Drug: Boceprevir, Peg-interferon alfa 2b and Ribavirin — * Screen period from Week-8
  * Standard treatment from day 0 to week 4 (W4)
  * Three-drug-regimen (Boceprevir introduction) from W4 to W8
  * HCV RNA determination at W8 determines treatment group and participation duration:
    * If undetectable HCV RNA at W8, it is a complete virological response: 3 drug-regimen is continued until W48, then there is a follow-up period up to W72 and SVR analysis,
    * If HCV RNA ≤ 1000IU/mL at W8, it is an incomplete virological response. The 3-drug-regimen is continued until W72, when another analysis is done.
  Other Names: ViraferonPeg; Rebetol

SUMMARY:
The majority of Human immunodeficiency Virus (HIV)/Hepatitis C Virus (HCV) co-infected patients are non responders after 48 weeks of the current standard-of-care with Peg-Interferon/Ribavirin. The results of re-treatment are disappointing. The addition of Boceprevir to the current standard-of-care has been shown to increase the efficacy of therapy in HCV mono-infected patients previously treated with a bi-therapy. Knowing that HIV/HCV co-infected patients are subject to more rapid hepatic fibrosis as well as to increased risks of cirrhosis, end-stage liver disease and hepatocellular carcinoma, it is important to improve the response rate of the re-treatment of hepatitis C in these patients.

The aim of this pilot study is to evaluate the efficacy and safety of Boceprevir in combination with Peg-Interferon alfa 2b plus ribavirin, in patients co-infected with HIV and chronic genotype 1 HCV, and previously treated with Peg-Interferon/Ribavirin. 80 subjects will be enrolled. The primary endpoint will be the Sustained Virologic Response (SVR) defined as undetectable HCV-RNA at Week 24 after the end of therapy.

DETAILED DESCRIPTION:
The majority of HIV/HCV co-infected patients are non responders after 48 weeks of the current standard-of-care with Peg-Interferon/Ribavirin. The results of re-treatment are disappointing. The addition of Boceprevir to the current standard-of-care has been shown to increase the efficacy of therapy in HCV mono-infected patients previously treated with a bi-therapy. Knowing that HIV/HCV co-infected patients are subject to more rapid hepatic fibrosis as well as to increased risks of cirrhosis, end-stage liver disease and hepatocellular carcinoma, it is important to improve the response rate of the re-treatment of hepatitis C in these patients.

Subjects enrolled in this trial will have many predictive factors of failure: HIV co-infection, previous failure to Peg-Interferon/Ribavirin, HCV genotype 1 infection. One study reported a SVR rate of 9% after re-treatment with Peg-Interferon/Ribavirin in such patients. Another trial has shown a substantial increase of the response rate with a tri-therapy in HCV mono-infected patients.

The investigators propose to carry out a multicentric, national, non-randomized phase II trial in 80 patients.

The proportion of patients with F4 cirrhosis will have to be inferior to 50% of enrolled subjects.

The number of null responders to a previous treatment (HCV RNA drop < 2 log10 at W12) and without F4 cirrhosis will have to be lower or equal to 20.

The primary objective of the study is to estimate, in Genotype 1 - HCV/HIV co-infected patients, non responders to a previous therapy with Peg-Interferon/Ribavirin, the rate of SVR after 48 or 72 weeks of a three-drug regimen containing Peg-Interferon, Ribavirin and Boceprevir according to the Virologic Response and to compare the SVR rate to a threshold rate 20%, lowest rate to consider a therapeutic benefit in this population.

A pharmacokinetic sub-study including 30 patients will be performed to estimate pharmacokinetic parameters of antiretroviral treatment (Atazanavir combined with Ritonavir, Raltegravir, Tenofovir) in combination with anti HCV treatment at baseline and W8 and pharmacokinetic parameters of Boceprevir at W8.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18 years
* HIV-1 infection
* Infection to genotype 1 HCV only
* Patients must have received at least 12 weeks of treatment with Peg-Interferon alfa 2a ≥ 135 µg / once weekly or Peg-Interferon alfa 2b ≥ 1,0 µg/kg/ once weekly + Ribavirin ≥ 600 mg daily and must have failed to treatment.
* Anti-HCV treatment stopped for at least 6 months
* Patients must be already treated at screen since at least 3 months with a stable combination of antiretroviral treatment as following:

  * Either tenofovir - emtricitabine, and atazanavir in combination with ritonavir
  * Or tenofovir - emtricitabine, and raltegravir
  * If patients cannot receive neither of the two antiretroviral regimens proposed, for virologic, safety or toxicity reasons, patients could receive any effective antiretroviral therapy including : tenofovir, emtricitabine, lamivudine, atazanavir alone or in combination with ritonavir, raltegravir, abacavir. These patients are not allowed to take part in the pharmacokinetic sub-study.
* CD4 > 200/mm3 et >15%, at screen
* HIV-RNA < 50 copies/ml since at least 6 months at screen
* ≥ 40 Kg and ≤ 125 Kg
* Patients with any fibrosis grade. Proportion of F4 subjects should not excess 50% of the overall subjects.
* Male and female subjects must agree to use acceptable methods of contraception 1 month prior to starting the study treatment and to continue until 7 months after the last doses of study drugs for male subjects and their partner(s), 4 months for female subjects.
* Subjects must be willing to give written informed consent for principal study (signed at least at screen visit and prior to any study investigation)and + for the pharmacokinetic sub-study (for the concerned centers).
* Subjects must be willing to give written informed consent for biological collection.
* Subjects must be willing to give written informed consent for treatment of genetics data.
* Subjects affiliated or beneficiary to a medical insurance.

Exclusion Criteria:

History:

* Patients with cirrhosis (F4) and nul responders to prior treatment
* Cirrhosis classified Child-Pugh B or C or history of decompensated cirrhosis of the liver. If Child A classification, significant varicose veins (grade 2 or 3) observed with a fibroscopy realized for < 3 years.
* History of ocular neuritis, retinal disorders, transplant
* Opportunistic infections (classification C), active or occurred within the 6 months prior to baseline.
* History of neoplasia within the last 5 years, except cutaneous basocellular carcinoma, recovering Kaposi's sarcoma, in situ cervical or anal canal cancer.

Current condition:

* Co-infection with Hepatitis B virus
* Pregnancy and lactation
* Cardiac or severe pulmonary disease
* Untreated dysthyroidism
* Autoimmune disease contraindicating to an interferon treatment
* Severe haemoglobinopathies
* Any condition needing a systemic corticotherapy or an immunosuppressive treatment
* Evolutive current malignancy, including hepatocarcinoma which should be specifically controlled prior to baseline.
* Alcohol consumption which may disturb the study participation according to the investigator
* Drug addiction which may disturb the study participation according to the investigator. Patients taking part to a substitution program with methadone or buprenorphine are allowed to be enrolled in the study.

Biological criteria:

• Haemoglobin < 12 g/dL (female) or < 13g/dL (male), Platelets < 90 000/mm3, Neutrophil count < 1500/mm3, Renal failure defined as creatinine clearance < 50ml/min, Uncontrolled thyroid function, HbA1c ≥ 7% in case of diabetes

Criteria related to study drugs

* Contra-indication to Ribavirin, interferon treatment including psychiatric contra-indications.
* History of discontinuation for intolerance to anti-HCV treatment.Patients with a history of discontinuation for intolerance, especially anaemia or leuconeutropenia, and who were not treated with hematopoietic growth factor, are eligible
* Concomitant medication which may interfere with Boceprevir, atazanavir, ritonavir and raltegravir pharmacokinetic
* St.John's-wort consumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Sustained Virologic Response | Week 72 or Week 96 (W72 or W96)
  HCV-RNA measured 24 weeks after the end of the HCV treatment (W72 or W96)

SECONDARY OUTCOMES:
HCV viral load | W4, W8, W12, W16, W28, W36 and at treatment completion at W48/72
  HCV-RNA
Predictive factors of Sustained virologic Response (SVR) | Baseline
  * Sex
  * Age (< vs ≥ 40 years)
  * Risk factor of HIV infection (drug consumer versus other risk factors)
  * Risk factor of HCV infection (drug consumer versus other risk factors)
  * Ethnic origin (Africano-American or Subsaharian-African or West Indies versus others)
  * CDC stade (C vs. A-B)
  * CD4 number (< vs. ≥ 350/mm3)
  * HCV viral load (< versus ≥ 800 000 UI/ml)
  * HCV genotype (1a versus 1b)
  * Cirrhosis (F4 versus no cirrhosis)
  * Alcohol, tobacco, cannabis, intravenous/nasal drugs consumption
  * IL28 gene polymorphism
HIV virologic endpoints | W4, W8, W12, W16, W20, W24, W28, W32, W36, W40, W44, W48, W60, W72 and W84, W96 if treatment duration is 72 weeks
  * HIV-RNA
  * CD4 and CD8 count
Residual plasmatic concentration (Cres) of Ribavirin | W4 and W8
Hepatic factors: liver fibrosis score | Screen, W4, W8, W16, W28, W48, W72, W96.
  Evolution of liver fibrosis between baseline and 24 weeks post-treatment, according to baseline value and Sustained Virologic Response (at W4, W8, W16, W28, W48/72 and 24 weeks post-treatment).
Alcohol consumption | W4, W8, W16, W28, W48, W72, W96
Evaluation of Pharmacokinetic parameters of anti-retroviral treatments | Day 0, W8
  Pharmacokinetic parameters (Cres, Cmax, AUC) of anti-retroviral treatments before (baseline) and after (W8) the starting of Boceprevir combination in a sub-group of subjects and according to UGTA1 polymorphism.
Clinical and biological adverse events | Up to 24 weeks after treatment completion (W72 or W96)
Number of participants classified by virologic failure type: non responder, relapser, null responder | W8, W12, W16, W28, W48, W72, W96
  * Relapse patients: undetectable HCV RNA at the end of therapy, becoming detectable after treatment cessation.
  * Break-through patients: undetectable HCV-RNA at least once during treatment, becoming detectable before treatment cessation.
  * Non-responder patients: detectable HCV-RNA at W24, never achieved undetectable and HCV RNA drop ≥ 2 log at W12.
  * Null responder patients: HCV RNA drop < 2 log at W12
ITPA gene polymorphism | Day 0
  The relation between ITPA gene polymorphism and onset of haemolytic anaemia will be analysed.
CYP3A4 Polymorphism | W8
  Evaluation of Pharmacokinetic parameters (Cres, Cmax, AUC) of Boceprevir at W8 in a sub-group of subjects, according to antiretroviral treatment and CYP3A4 polymorphism.
Maximal Concentration (Cmax) of antiretroviral treatments | Day 0 and W8
  Evaluation of Pharmacokinetic parameters (Cres, Cmax, AUC) of anti-retroviral treatments before (baseline) and after (W8) the starting of Boceprevir combination in a sub-group of subjects and according to UGTA1 polymorphism.
Area Under the Curve (AUC) of antiretrovirals | Day 0 and W8
  Evaluation of pharmacokinetic parameters (Cres, Cmax, AUC) of anti-retroviral treatments before (baseline) and after (W8) the starting of Boceprevir combination in a sub-group of subjects and according to UGTA1 polymorphism.
Insulin resistance | at W4, W8, W16, W28, W48, W72, W96
  Evolution of insulin resistance between baseline and 24 weeks post-treatment according to baseline value and Sustained Virologic Response (at W4, W8, W16, W28, W48/72 and 24 weeks post-treatment).
Metabolic syndrome | W4, W8, W16, W28, W48, W72, W96
  Evaluation of metabolic syndroms parameters according to baseline value and Sustained Virologic Response (at W4, W8, W16, W28, W48/72 and 24 weeks post-treatment).
Reasons and dates of treatment discontinuation | Up to W72
Perceived symptoms | Day 0, W28, W48, W72, W96
  Perceived symptoms will be assessed on "AC24 French AIDS scale"
French AIDS questionnaire of compliance | W0, W28, W48, W72
Tobacco consumption | W4, W8, W16, W28, W48, W72, W96
Cannabis consumption | W4, W8, W16, W28, W48, W72, W96
Intravenous/nasal drugs consumption | W4, W8, W16, W28, W48, W72, W96
Residual Concentration (Cres) of atazanavir boosted or not by ritonavir | At screening day, at W48 and in the case of virological rebound
  Measure of residual concentration of atazanavir for patients treated by atazanavir boosted or not by ritonavir at screening day, at W48 and in case of virological rebound (HIV and HCV).
Residual concentration (Cres) of ritonavir | At screening day, at W48 and in the case of virological rebound
  Measure of residual concentration of ritonavir for patients treated by atazanavir boosted by ritonavir at screening day, at W48 and in case of virological rebound (HIV and HCV).

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Poizot-Martin, MD, Principal Investigator — University Hospital, Marseille; Eric Bellissant, MD, PhD, Study Chair — Rennes University Hospital
Locations (1):
- CHU Sainte Marguerite, Marseille, France

REFERENCES:
- [Derived] Poizot-Martin I, Bellissant E, Garraffo R, Colson P, Piroth L, Solas C, Renault A, Bourliere M, Halfon P, Ghosn J, Alric L, Naqvi A, Carrieri P, Molina JM; ANRS HC27 BOCEPREVIH Study Group. Addition of boceprevir to PEG-interferon/ribavirin in HIV-HCV-Genotype-1-coinfected, treatment-experienced patients: efficacy, safety, and pharmacokinetics data from the ANRS HC27 study. HIV Clin Trials. 2016 Mar;17(2):63-71. doi: 10.1080/15284336.2015.1135553. Epub 2016 Feb 11. PMID 27077673